#### STATISTICAL ANALYSIS PLAN

Study Code

D589BC00027

Edition Number 4.0

Date

29-Jul-2024

# **CARE FOR ALL**

Change Asthma Clinical Practice through Guideline Education and Implementation For All Patients with Asthma: an **Evaluation of an Asthma Quality Improvement Program** 

# TABLE OF CONTENTS

| TITLE PAG | 3E | . 1 |
|----------------|---------------------------------------------------|-----|
| TITLE PAG | GE | . 2 |
| TITLE PAG | GE | . 3 |
| TITLE PAG | GE | . 4 |
| TABLE OF | CONTENTS | . 5 |
| LIST OF A | BBREVIATIONS | . 7 |
| AMENDM | ENT HISTORY | . 8 |
| 1 | INTRODUCTION | 11 |
| 1.1 | Study Objectives | 11 |
| 1.2 | Study Design | 14 |
| 1.3 | Number of Subjects | 20 |
| 2 | CHANGES TO PROTOCOL PLANNED ANALYSES | 20 |
| 3 | DATA ANALYSIS CONSIDERATIONS | 20 |
| 3.1 | General Considerations | 20 |
| 3.1.1 | General Study Level Definitions | |
| 3.1.2 | Baseline Definition | |
| 3.1.3 | Study Day | |
| 3.1.4 | Visit Window | |
| 3.1.5 | Handling of Unscheduled Visits | |
| 3.1.6 | Handling of Protocol Deviations in Study Analysis | 22 |
| 3.1.7 | Handling of Missing Data | |
| 4 · | STATISTICAL ANALYSIS | |
| 4.1 | Study Population | |
| 4.1.1 | Subject Disposition and Completion Status | |
| 4.1.2 | Analysis Sets | |
| 4.1.3 | Protocol Deviation | |
| 4.1.4 | Demographics | |
| 4.1.5<br>4.1.6 | Disease Characteristics | |
| 4.1.7 | Medical History and Concomitant Disease | |
| 4.1.8 | Prior and Concomitant Medications | |
| 4.1.9 | Prescriptions | |
| 4.2 | Endpoint Analyses | |
| 4.2.1 | Primary Endpoint | |
| 4.2.1.1 | Definition | |
| 4.2.1.2 | Primary Analysis of Primary Endpoint | |
| 4.2.1.3 | Sensitivity Analyses of the Primary Endpoint | |
| 4.2.1.4 | Supplementary Analyses of the Primary Endpoint | |
| 4.2.2 | Secondary Endpoints | 27 |

| STATISTICA | AL ANALYSIS PLAN | AstraZeneca |
|---|---|---|
| D589BC0002 | 27 – ed.4.0 | 29-Jul-2024 |
| 4.2.2.1 | Secondary Endpoint-1 | 27 |
| 4.2.2.2 | Secondary Endpoint-2 | 28 |
| 4.2.2.3 | Secondary Endpoint-3 | |
| 4.2.2.4 | Secondary Endpoint-4 | 28 |
| 4.2.2.5 | Secondary Endpoint-5 | |
| 4.2.3 | Other Endpoint | 29 |
| 4.2.3.1 | Exploratory Endpoint-1 | 29 |
| 4.2.3.2 | Exploratory Endpoint-2 | |
| 4.2.3.3 | Exploratory Endpoint-3 | 30 |
| 4.2.3.4 | Exploratory Endpoint-4 | 30 |
| 4.2.3.5 | Exploratory Endpoint-5 | 31 |
| 4.2.3.6 | Exploratory Endpoint-6 | |
| 4.2.3.7 | Exploratory Endpoint-7 | |
| 4.2.3.8 | Exploratory Endpoint-8 | |
| 4.2.3.9 | Exploratory Endpoint-9 | 33 |
| 4.2.3.10 | Exploratory Endpoint-10 | |
| 4.2.3.11 | Exploratory Endpoint-11 | |
| 4.2.3.12 | Exploratory Endpoint-12 | |
| 4.2.3.13 | Exploratory endpoint-13 | |
| 4.2.4 | Subgroup analyses | 35 |
| 5 | INTERIM ANALYSIS | 37 |
| 6 | REFERENCES | 39 |
| 7 | APPENDIX | 40 |
| 7.1 | SAS sample code for proc GLIMMIX | |
| 7.2 | SAS sample code for proc GENMODE | 40 |
| 7.3 | ASTHMA QUALITY OF LIFE QUESTIONNAIRE WITH STANDARDISED ACTIVITIES (AQLQ(S)) | 40 |

# LIST OF ABBREVIATIONS

List abbreviations and definitions of specialized or unusual terms, measurements, or units. Examples are provided below. These can be modified at study level.

| Abbreviation or<br>Specialized<br>Term | Definition |
|---|---|
| AE | Adverse Event |
| BPT | Bronchial Provocation Test |
| CRO | Contract Research Organisation |
| CSP | Clinical Study Protocol |
| CSR | Clinical Study Report |
| eCRF | electronic Case Report Form |
| FeNO | Fractional exhaled Nitric Oxide |
| GCP | Good Clinical Practice |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IMP | Investigational Medicinal Product |
| IRB | Institutional Review Board |
| KPI | Key Performance Indicator |
| MCID | Minimum Clinical Important Difference |
| PEF | Peak Expiratory Flow |
| PFT | Pulmonary Function Testing |
| PHL | Potential Hy's Law |
| PI | Principal Investigator |
| QIP | Quality Improvement Program |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SoA | Schedule of Activities |

# AMENDMENT HISTORY

| CATEGORY Change refers to: | Date | Description of change | In line with CSP? | Rationale |
|---|---|---|---|---|
| N/A | 10/21/2022 | Initial approved SAP | Yes | N/A |
| N/A | 7/4/2022 | Add 2 interim analysis per<br>Protocol v2.0 | Yes | N/A |
| Exploratory<br>Endpoints | 7/4/2023 | Add below exploratory endpoints per Protocol v2.0- | Yes | N/A |
| | | 1 | | |
| | | - a 3 <sub>1</sub> | · s | |
| | | • | | |
| | | • | | |

| CATEGORY Change refers to: | Date Description of change | | In line with CSP? | Rationale |
|---|---|---|---|---|
| В | | characteristic and asthma control level | | |
| N/A 2/18/2024 window for investigator analysis. | | Add scope of the interim | Yes | N/A |
| Exploratory<br>Endpoints | 2/18/2024 | Add below exploratory endpoints per protocol V3.0 | Yes | N/A |
| NA Specify the visit windowing strategy for investigators in details, similar to subject's windows rule. | | Yes | N/A | |
| Subgroup Anlyses | 8/19/2024 | Move all subgroup analyses to a separate section 4.2.4. Specify the definition and cut-off threshold for subgroups. | Yes | N/A |
| Exploratory<br>Endpoints - 3 | 8/19/2024 | | Yes | N/A |
| Exploratory<br>Endpoints -5 | 8/19/2024 | | No | Prior and concomitant medication page does not collect the investigator ID number, so deleted. |
| NA | 8/19/2024 | Change wording "partially controlled" to "partly controlled" for ACQ-5 (0.75 to 1.5). | No | Based on<br>comments from<br>expert opinion, the<br>word "partially" is |

| CATEGORY Change refers to: | Date | Description of change | In line with CSP? | Rationale |
|---|---|---|---|---|
| | | | | not correct for ACQ-5 (0.75 to 1.5), so changed to "partly". |
| Safety analyses | 8/19/2024 | Deleted safety analysis part<br>to be consistent with CSP<br>V3.0 (with no safety<br>objective or endpoints in<br>CSP) | Yes | N/A |

## 1 INTRODUCTION

This statistical analysis plan is for AstraZeneca "Change Asthma Clinical Practice through Guideline Education and Implementation For All Patients with Asthma: an Evaluation of an Asthma Quality Improvement Program (short title: CARE FOR ALL: an Evaluation of an asthma QIP)" (Study code: D589BC00027) and will give a detailed description of it. This version of SAP is for final analysis plan.

This is a real-world, multi-centre prospective study to bridge the gap that exists between GINA guideline recommendations and current clinical practice by demonstrating the benefits of an asthma quality improvement program (QIP), i.e. a standardized pulmonologist-targeted GINA guideline education and practice implementation. This is an evaluation on an asthma Quality Improvement Program (QIP, including GINA guideline education/training and implementation) to understand the change of physician behaviours, which leads to the change of patient outcomes.

This statistical analysis plan is based on the 3.0 version of the research protocol on February 22, 2023, the 5.0 version of the Case Report Form on September 26, 2023.

# 1.1 Study Objectives

| Ob | jectives | Endpoints |
|---|---|---|
| Pri | mary | |
| • | To evaluate the change in GINA guideline-<br>recommended treatments after guideline<br>education and implementation. | Change from baseline in the proportion of participants with an ICS-based maintenance and/or reliever treatment at week 48 |
| Sec | ondary | |
| • | To describe the asthma control after guideline education and implementation. | Secondary Endpoint 1 Change from baseline in the proportion of participant with well-controlled asthma (ACQ-5 ≤ 0.75) at week 48 |
| | | <ul> <li>Distribution of ACQ-5 average scores [proportion of subjects well-controlled (ACQ-5 ≤ 0.75), partly controlled (0.75 to 1.5) and not well-controlled (ACQ-5 ≥ 1.5)] at weeks 12, 24, 36 and 48 </li> </ul> |
| • | To describe the change in GINA guideline-<br>preferred treatments during guideline<br>education and implementation. | Secondary Endpoint 2 Change from baseline in the proportion of participants on the treatment of ICS-formoterol as reliever at week 12, 24, 36 and 48 |
| • | To describe the change in asthma control during guideline education and implementation. | Secondary Endpoint 3 Change from baseline in ACQ-5 average score at week 12, 24, 36 and 48 |
| | | Change from baseline in the proportion of participants achieving an improvement in ACQ-5 MCID of 0.5 units or more at week 12, 24, 36 and 48 |
| • | To describe the change in GINA guideline-<br>recommended treatments during guideline<br>education and implementation. | Secondary Endpoint 4 Change from baseline in the proportion of participants with an ICS-based maintenance and/or reliever treatment at week 12, 24 and 36 |
| • | To describe asthma related treatment patterns during the study duration. | Secondary Endpoint 5 Asthma related treatment patterns - Asthma treatment distribution at baseline and weeks 12, 24, 36, and 48, e.g., ICS-containing medications, ICS-LABA, ICS-formoterol, oral corticosteroids, leukotriene receptor antagonists, |

| | theophylline, Traditional Chinese |
|-------------|-----------------------------------|
| | Medicine |
| Exploratory | |
| • | |
| | • |
| • | |
| • | |
| • | |
| • | |
| • | |
| - | |
| • | _ |
| • | |
| _ | |
| • | |

| • | |
|---|---------|
| • | - + 1 1 |
| • | |

# 1.2 Study Design

The study will select a total of around 30 Tier 2 and Tier 3 hospitals across China and enrol approximately 1500 asthma patients ≥14 years old with all severities from the 30 participating hospitals. To represent the real-world situation of patients, pulmonologists and treatment practice, hospital selection will include as many as provinces or municipalities in mainland China, where the altitude is below 1,500 meters, while balancing hospital grade (e.g. 10 Tier 2 and 20 Tier 3). Patients will be recruited in hospital outpatient setting, where all potentially eligible asthma patients will be consecutively approached and invited to join the study, e.g., regardless of new patients or treated, exacerbation or regular follow-up.

The QIP (i.e., GINA 2021 guideline education/training and implementation) will be delivered to pulmonologists and specialist nurses in participating hospitals at hospital level, including pulmonologist-targeted initial comprehensive education based on GINA 2021, guideline implementation performance assessment and feedback, reinforcement learning, along with multiple online and offline approaches serving as reminders and supportive tools to ensure consistent education and to facilitate the asthma management in daily clinical practice in accordance with GINA 2021 recommendation.

Immediately after last patient has been enrolled at each site, the study intervention will be initiated, i.e., the initial comprehensive training on GINA 2021 will be offered to pulmonologists and specialist nurses in this hospital. All successfully enrolled participating patients will be followed up for up to 48 weeks and return to recruiting hospital for study

visits every 12 weeks. The total participating duration in this study for each participating patient will be approximately 60 weeks.

The study aims to bridge the gap between the recommendations from GINA 2021 and current clinical practice via an asthma QIP (including GINA guideline education/training and implementation).



**Table 1 Schedule of Activities (participating patients related)** 

| | Baseline<br>Period | | Intervention Period | | | Details in CSP<br>Section or Appendix | |
|---|---|---|---|---|---|---|---|
| Study Visit | Vo | V1 | V2 | V3 | V4 | V5<br>(Study completion/<br>withdrawal) | |
| Weeks | -12<br>±7 | 0<br>±<br>14 | 12<br>±7 | 24<br>±7 | 36<br>±7 | 48<br>±7 | |
| Informed consent a | Х | | | | | | |
| Inclusion and exclusion criteria | х | | | | | | Sections 5.2.1 and 5.2.2 |
| Demographics <sup>b</sup> | Х | | | | | | |
| Vital Sign <sup>c</sup> | X | | | | | | |
| Subject status <sup>d</sup> | X | | | | | | |
| Smoking status <sup>e</sup> | X | | | | , | | |
| Medical history (comorbidities) and medications f | X | | | | | | |
| Asthma history & related treatment <sup>g</sup> | Х | | | | | | |
| Severe asthma exacerbation | | х | Х | Х | Х | Х | |
| Hospitalization due to asthma exacerbation since last visit | | Х | Х | Х | Х | Х | Section 8.1.4 |
| ACQ-5 | X | Х | Х | Х | Х | X | Section 8.1.5.1 |
| AQLQ(S)+12 | X | Х | Х | Х | X | X | Section 8.1.5.2 |
| PFT | Х | | | | | X | |
| MARS-A questionnaire | X | | Х | Х | | Х | |
| Questionnaire of asthma knowledge for patient | X | | Х | Х | | X | |
| Inhale skill score for patient | | Х | Х | X | | Х | |
| Patient's expectation for asthma treatment | Х | | Х | Х | | х | |

| | Baseline<br>Period | | | Interv | Intervention Period | Period | Details in CSP<br>Section or Appendix |
|---|---|---|---|---|---|---|---|
| Study Visit | 0A | N1 | 42 | V3 | V4 | V5<br>(Study completion/<br>withdrawal) | |
| Laboratory assessments within prior 3 months (if available in medical records) h | × | × | × | × | X | X | |
| PFT/BPT/PEF/FeNO within prior 3 months (if available in medical records) | × | X | × | X | X | X | |
| Medical records on asthma related assessment and treatment | × | Х | × | Х | Х | X | |
| Questionnaire for Asthma Patients during COVID-19i | | | i | X | | | Section 8.1.9 |
| Patient evaluation on whose pulmonologists 1. assess symptom control, 2. watch the patient using their inhaler, educate their technique, 3. have a discussion about adherence, 4. develop or review the written asthma action plan, provide patient education, 5. had a PFT before dosage reduction | × | × | × | × | × | × | Section 6.1.2.3 |

PFT = Pulmonary Function Testing, BPT = Bronchial provocation test, PEF = Peak expiratory flow, FeNO = Fractional exhaled nitric oxide

- a. Informed consent must be conducted prior to performing any study procedures including data collection.
- b. Demographic includes patient age, gender, race, ethnicity and
- c. Vital signs include body mass index (BMI, calculation by height and weight)
- d. Subject Status education level, family monthly income, job, residence (urban communities or rural villages), etc
  - e. Smoking status include current smoker or stopping smoking or restarting smoking, smoking pack-years
- f. Asthma related comorbidities, including allergic history, rhinitis, chronic rhinosinusitis, nasosinusitis, gastroesophageal reflux disease, obesity, obstructive sleep apnea, depression, anxiety, eczema, and atopic dermatitis according to ICD-10-CM.Medication includes drugs administered for these asthma related comorbidities within 4 weeks before enrolment
- g. Historical data, e.g., the first diagnosed date of asthma and total asthma exacerbation, total number of prescription of systemic glucocorticoid treatment for at least 3 days or emergence visit or hospitalization due to asthma exacerbations during previous 12 months (an emergency room visit due to asthma that required use of systemic corticosteroids or hospitalization due to asthma), home PEF availability, asthma symptoms, severity class evaluated by self-assessment, asthma control level, first asthma-diagnose hospital and Tiers level, hospital numbers for asthma clinic visit in past 12month, medical insurance category, Patient's expectation for asthma treatment, etc
- h. Clinical laboratory testing data include CBC with differentiation, blood gas analysis (pH, SaO2, PaO2, PaCO2, and HCO3-); C-reactive protein; skin allegen prick, total IgE or specific IgE

i: If the patient got COVID-19 infection, then answer the questionnaire, the uninfected patients are not necessary to response. Every subject if has a new infected with COVID-19 should answer one time.

# 1.3 Number of Subjects

Approximately 1500 participants will provide 80% power at a significant level of 0.05 to detect a change from baseline in the proportion of patients with an ICS-based maintenance and/or reliever treatment at week 48 of 5%. The baseline proportion is assumed to be 40% and a within-participants correlation is assumed to be 0.25. The proportion of missing postbaseline assessment at week 48 is assumed to be 30%.

# 2 CHANGES TO PROTOCOL PLANNED ANALYSES

Not Applicable

## 3 DATA ANALYSIS CONSIDERATIONS

## 3.1 General Considerations

Unless otherwise stated, all statistical methods in the subsequent sections will be based on the following general methods. Statistical programming and analyses will be performed using SAS® (SAS Institute, Inc., Cary, NC, USA), version 9.3 or higher, and/or other validated statistical software as required

All categorical data will be presented in contingency tables, using absolute and relative frequencies. Percentages will be rounded to the first decimal place and, therefore, may not always add up to 100%. When applicable, 95% confidence intervals (CIs) will be presented with estimates of proportions. The percentages will not be presented for zero counts.

All continuous data will be summarized via relevant descriptive statistics, such as number of observations with available measurements, mean, standard deviation, median, first and third quartiles (Q1 and Q3) when applicable, minimum and maximum.

Missingness in the variables will also be presented.

Decimal points will be presented as follows: N will be presented without decimal, minimum/maximum in same precision as in the database, mean/median in one more decimal than minimum/maximum, and SD in one more decimal than mean/median. And the decimal places of SD should not be greater than 4.

## 3.1.1 General Study Level Definitions

The Electronic Data Capture (EDC) system will be used for data collection and query handling. Except for the questionnaires to be completed by participants, all data will be based on what have been generated during routine clinical practice, if available.

## 3.1.2 Baseline Definition

Unless otherwise stated, general baseline will be defined as the last non-missing evaluation on or prior to Visit 0. Baseline definitions of comorbidities and treatments are provided in the comorbidities, medications and prescriptions sections (refer to section 4.1.8 and 4.1.9).

## 3.1.3 Study Day

If the assessment date is on or after Visit 1 in intervention period, the study day will be calculated as: Assessment Date – Date of Visit 1 in intervention period + 1.

If the assessment or event date is prior to Visit 1 in intervention period, the study day will be calculated as: Assessment Date – Date of Visit 1 in intervention period.

#### 3.1.4 Visit Window

A visit windowing strategy will be implemented for subjects as shown below.

| Analysis visit | Target Day | Actual assessment day |
|----------------|------------|-----------------------|
| Week 0 | Day 1 | Training day to D42 |
| Week 12 | Day 84 | D43 to D126 |
| Week 24 | Day 168 | D127 to D210 |
| Week 36 | Day 254 | D211 to D294 |
| Week 48 | Day 336 | D295 to D378 |

The visit will be missing if no assessment was reported within the specified visit window. If multiple assessments fall within one visit window, the scheduled visit takes priority, followed by the one closest to the target day. If two evaluations are equidistant from the scheduled time point, the earlier one will be used.

A visit windowing strategy will be implemented for investigator as shown below:

| Analysis visit | Target Day | Actual assessment day |
|----------------|------------|-----------------------|
| Baseline | | <= Training day |
| Week 12 | Day 84 | Day2 to D126 |
| Week 24 | Day 168 | D127 to D252 |

| Week 48 | Day 336 | D253 to D378 |
|---------|---------|--------------|

The visit will be missing if no assessment was reported within the specified visit window. If multiple assessments fall within one visit window, the one closest to the target day. If two evaluations are equidistant from the scheduled time point, the earlier one will be used.

# 3.1.5 Handling of Unscheduled Visits

Listings will include scheduled and unscheduled data.

## 3.1.6 Handling of Protocol Deviations in Study Analysis

Criteria for protocol deviations will be established, and patients with protocol deviations will be identified and documented before the database lock.

## 3.1.7 Handling of Missing Data

Missing data will not be imputed unless otherwise specified elsewhere in the SAP.

Missing dates or partially missing dates will be imputed conservatively for adverse events and prior or concomitant medications/procedures.

For comorbidities, medications and prescriptions sections, incomplete (i.e., partial missing) date will be imputed.

#### **Incomplete End Date:**

If missing day and month, then December 31 will be assigned to the missing field.

If missing day only, then the last day of month will be assigned to the missing field.

If the death date is complete and the imputed end date is after the death date, then the end date will be imputed using the death date.

## Incomplete Start Date/Baseline Prescribed Date

If missing day and month, then January 1 will be assigned to the missing field.

If missing day only, then the first day of month will be assigned to the missing field.

If the imputed start date is after the end date, then the start date will be imputed using the end date.

If the imputed baseline prescribed date is after the planned start date, then the baseline prescribed date will be imputed using the planned start date.

Otherwise, do not impute.

For incomplete asthma symptoms start date or asthma diagnosed date, the imputation will follow as below:

If missing day and month, then January 1 will be assigned to the missing field.

If missing day only, then the first day of month will be assigned to the missing field.

Otherwise, do not impute.

By-visit endpoints will be analyzed using observed data, unless otherwise specified. For observed data analyses, missing data will not be imputed and only the observed records will be included.

#### 4 STATISTICAL ANALYSIS

This section provides information on definitions, derivation and analysis/data presentation per domain.

# 4.1 Study Population

The domain study population covers subject disposition, analysis sets, protocol deviations, demographics, baseline characteristics, medical history and prior and concomitant medication.

## 4.1.1 Subject Disposition and Completion Status

The number of subjects who signed the informed consent will be calculated.

The number and percentage of subjects who enrolled, completed the study, remained on study and withdrew early will be summarized. The number and percentage of subjects who withdrew early for various reasons will be summarized according to the categories in the CRF. Study follow-up time and primary reason for screen failure will be summarized. Listing will also be presented.

Study Follow-up Time = EOS – training date +1

## 4.1.2 Analysis Sets

Effectiveness analyses will be performed using an FAS population. Demographic and baseline characteristics will be presented for both all participants analysis set and FAS. The following populations are defined:

All Enrolled Participants Analysis Set: All participating patients enrolled for the study without screen failure will be included in the All Enrolled Participants population.

Full Analysis Set (FAS): All enrolled participants with at least one non-missing post-intervention GINA guideline treatment assessment.

Based on all enrolled subjects, the number and percentage of subjects in the FAS will be calculated and summarized. Listing will be provided for the reason of exclusion from analysis sets.

#### 4.1.3 Protocol Deviation

Major protocol deviations will be summarized for all patients in FAS. They will also be listed by each category. No patients will be excluded from analysis from the FAS due to protocol deviations.

#### 4.1.4 Demographics

Demographics will be summarized using descriptive statistics for both all enrolled participants analysis set and FAS.

Continuous demographic variables include age, weight, height, and BMI (in kg/m²); categorical variables include age group (>65 years, ≥18 to ≤65 years, <18 years), sex, race, ethnicity, BMI group (≥24 kg/m², <24 kg/m²), education level, household per capita monthly income, occupation, residence, and source of drug purchase.

#### 4.1.5 Baseline Characteristics

Baseline characteristics will be summarized using descriptive statistics for both all enrolled participants analysis set and FAS.

Continuous baseline variables include number of pack years (current usage only); categorical variables include nicotine usage frequency (current, former, never), temporarily stop nicotine use for more than 6 months (current usage only).

#### 4.1.6 Disease Characteristics

Disease characteristics will be summarized using descriptive statistics for both all enrolled participants analysis set and FAS.

Disease characteristics includes Asthma history and Historical asthma exacerbation.

Continuous Asthma history variables include asthma duration since symptom start, asthma duration since diagnosed and hospital numbers for asthma clinic visit in past 12 months; categorical variables include SABA usage within one year before enrolment, Allergen Asthma Trigger, Any symptoms within the past 12 months, Most frequent symptoms within past 12 months and other symptom related questions in Asthma history CRF page.

Asthma duration since symptom start (in months) = (ICF date – asthma symptoms start date +1)/365.25\*12

Asthma duration since diagnosed (in months) = (ICF date – asthma diagnosed date +1)/365.25\*12

Continuous Historical asthma exacerbation variables include Historical Asthma Exacerbation number, number of exacerbations resulted in emergency room treatment, number of exacerbations resulted in hospitalization, medication number; categorical variables include Historical Asthma Exacerbation to Record within the past 12 months.

A subject data listing of disease characteristics will be provided.

## 4.1.7 Medical History and Concomitant Disease

Respiratory Medical History (Comorbidities) will be coded using MedDRA codes of the version currently in effect at the time of database lock. The number (percentage) of patients reporting a history of any medical condition, as recorded on the CRF, will be summarized by system organ class and preferred term in FAS. A listing of respiratory medical history will be provided.

## 4.1.8 Prior and Concomitant Medications

Prior and concomitant medications for asthma, and prior medications for asthma related comorbidities will be coded using the World Health Organization Drug Dictionary (WHO DD) of the version currently in effect at the time of database lock. The number and percentage of patients who took prior and concomitant medications for asthma, prior medications for asthma related comorbidities will be summarized respectively by ATC medication class 2 and WHO DD preferred term (PT) in the FAS. Prior and concomitant medications will also be presented in a listing.

Prior medications are defined as those medications with an end date prior to enrolment. Concomitant medications are defined as those medications which are taken on or after Visit 1 (Week 0). This includes medications which start prior to Week 0 but continue after Week 0. Multiple drug usage in the same classification and preferred term by a subject will be counted only once.

#### 4.1.9 Prescriptions

Prescribed medication for asthma will be coded using the World Health Organization Drug Dictionary (WHO DD) of the version currently in effect at the time of database lock. The number and percentage of patients who are prescribed for asthma will be summarized respectively by ATC medication class 2 and WHO DD preferred term (PT) and visit in the FAS. Prescriptions will also be presented in a listing.

If treatment is prescribed at least once within 3months before Visit 0 (week -12), the subjects will be regarded as receiving this treatment at baseline. For Visit 2 (week 12), if treatment is prescribed at least once on or after Visit 1 and on or before Visit 2, the subjects will be regarded as receiving treatment at this visit. For Visit 3 -Visit 5 (week 24, 36 and 48), if treatment is prescribed at least once after last visit and on or before this visit, the subjects will be regarded as receiving treatment at this visit.

# 4.2 Endpoint Analyses

This section covers details related to the endpoint analyses such as primary, secondary, other endpoints including sensitivity and supportive analyses.

# 4.2.1 Primary Endpoint

#### 4.2.1.1 Definition

The primary endpoint is the proportion of patients with an ICS-based maintenance and/or reliever treatment, which is indicated by whether or not the treatment option includes ICS-containing medication. Change from baseline in the proportion of patients with an ICS-based maintenance and/or reliever treatment at week 48 will be analysed.

Doctor's prescription will be used to define this endpoint. The baseline and following analysis visits' definitions refer to section 4.1.9.

# 4.2.1.2 Primary Analysis of Primary Endpoint

Proportion of patients with an ICS-based maintenance and/or reliever treatment will be described using the frequency with ICS and corresponding percentage at baseline and week 48.

The primary analysis will use mixed effect logistic regression model, taking the measurement timepoint (baseline/post-baseline) as the fixed effect, hospital, pulmonologist and patient as the random effects. Logit link function will be used, and the model parameters will be estimated by maximum likelihood approach. The compound-symmetry variance-covariance structure will be used. In case of lack of convergency, hospital and prescriber factors will be removed from the model.

Within the framework of this model, first predict for all patients the probability of ICS usage at baseline/ post-baseline and then take the average over baseline/ post-baseline patients to get an estimate of proportion, and finally take the difference between the two proportions as the risk difference estimate, the 95% confidence interval of risk difference in proportion by bootstrapping method will be estimated and presented. Besides, Odds Ratio and P value from the model will also be estimated and presented. The analysis will be performed in FAS. Reference SAS code is shown in section 7.

If medication is taken at least once within 3 months before Visit 0 (week -12), the patients will be regarded as taking this medication at baseline. For Visit 2 (week 12), if medication is taken at least once on or after Visit 1 and on or before Visit 2 (within 3 months before this visit), the subjects will be regarded as taking medications at this visit. For Visit 3 -Visit 5 (week 24, 36 and 48), if medication is taken at least once after last visit and on or before this visit (within 3 months before this visit), the subjects will be regarded as taking medication at this visit.

# 4.2.1.3 Sensitivity Analyses of the Primary Endpoint

Sensitivity analysis will be conducted with generalized estimating equations (GEE) model using measurement timepoint (baseline/post-baseline) as the fixed effect, and subject ID is used to identify individual subjects. Reference SAS code is shown in section 7. Logit link function will be used for binary distribution. The model parameters are estimated by generalized estimating equations. Compound-symmetry working correlation matrix will be used to model the correlation of the responses from subjects.

# **4.2.1.4** Supplementary Analyses of the Primary Endpoint Not applicable.

# 4.2.2 Secondary Endpoints

# 4.2.2.1 Secondary Endpoint-1

The ACQ-5 is a shortened version of the full 7-item ACQ (Juniper et al 1999) that assesses asthma symptoms (night-time awakening, symptoms on awakening, activity limitation, shortness of breath, and wheezing) but omits the FEV1 measurement and SABA use from the original ACQ assessment. Patients are asked to recall how their asthma has been during the previous week by responding to 5 symptom questions. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-5 score is the mean of the responses. Mean scores of ≤0.75 indicate well controlled asthma, scores between >0.75 and <1.5 indicate partly controlled asthma, and a score ≥1.5 indicates not well controlled asthma (Juniper et al 2006). Individual changes of ≥0.5 are considered to be clinically meaningful (Juniper et al 2005).

The change from baseline in the proportion of well-controlled asthma evaluated by ACQ-5 score at week 48 will be derived using the percentage of patients with ACQ-5 score  $\leq$  0.75, its 95% confidence interval (95% CI) will be summarized descriptively. Normal approximation method will be used to calculate 95% CI.

Distribution of ACQ-5 average scores at baseline and weeks 12, 24, 36 and 48 will be described as summary and listing, using the frequency and percentage at each category listed below, a shift table will also be generated:

Well controlled: ACQ-5 ≤ 0.75

Partly controlled: 0.75 <ACQ-5< 1.5</li>

Not well-controlled: ACQ-5 ≥ 1.5

## 4.2.2.2 Secondary Endpoint-2

One secondary endpoint is the proportion of patients on the treatment of ICS-formoterol as reliever, without concomitant SABA. Change from baseline in the proportion of patients on the treatment of ICS-formoterol as reliever at week 12, 24, 36 and 48 will be summarized with its 95% confidence interval (95% CI). Normal approximation method will be used to calculate 95% CI. Doctor's prescription will be used to define this endpoint. The baseline and following analysis visits' definitions refer to section 4.1.9.

#### 4.2.2.3 Secondary Endpoint-3

The ACQ-5 overall score will be calculated as the average of the non-missing 5 symptom questions. At least 4 out of the 5 symptom items are needed to provide an ACQ-5 overall score. Change from baseline in ACQ-5 average score at week 12, 24, 36 and 48 will be summarized.

Responder status will be descriptively summarized by visit as the number (%) of responders and non-responders. A responder status at post-baseline will be calculated as

- Responder: (post-baseline baseline) ≤ -0.5
- Non-responder: (post-baseline baseline) > -0.5

Proportion of participants achieving an improvement in ACQ-5 MCID of 0.5 units or more at Week 12, 24, 36 and 48 will be summarized.

#### 4.2.2.4 Secondary Endpoint-4

Change from baseline in the proportion of patients with an ICS-based maintenance and/or reliever treatment at week 12, 24 and 36 will be summarized with its 95% confidence interval (95% CI). Normal approximation method will be used to calculate 95% CI.

## 4.2.2.5 Secondary Endpoint-5

Asthma related treatment patterns will be evaluated by treatment distribution at baseline and at weeks of 12, 24, 36 and 48, e.g., ICS-containing medications, ICS-LABA, SABA, ICS-formoterol, oral corticosteroids, leukotriene receptor antagonists, theophylline, Traditional Chinese Medicine and combination.

- 4.2.3 Other Endpoint
- 4.2.3.1 Exploratory Endpoint-1
- 4.2.3.2 Exploratory Endpoint-2

- 4.2.3.3 Exploratory Endpoint-3
- 4.2.3.4 Exploratory Endpoint-4

## 4.2.3.5 Exploratory Endpoint-5

## 4.2.3.6 Exploratory Endpoint-6

4.2.3.7 Exploratory Endpoint-7

# 4.2.3.8 Exploratory Endpoint-8

4.2.3.9 Exploratory Endpoint-9

- 4.2.3.10 Exploratory Endpoint-10
- 4.2.3.11 **Exploratory Endpoint-11**
- 4.2.3.12 Exploratory Endpoint-12

## 4.2.3.13 Exploratory endpoint-13

# 4.2.4 Subgroup analyses

Subgroup analyses as below will be performed as appropriate for the primary endpoint, selected secondary endpoints and exploratory endpoints. Any subjects with a missing value for the defined subgroup will be excluded from the analysis of that subgroup. The subgroups to be explored may include as needed:

- Age be category: >65 years, ≥18 to ≤65 years, <18 years old
- Age of onset: <20 years old, <40 years old, ≥40 years old
- Phenotype of asthma: allergic or non-allergic
- Hospital Tier: Tier 2, Tier 3
- Job: related to asthma, no-related to asthma (occupational exposure Y or N)
- Nicotine usage frequency (current, former, never)
- Sex (Male, Female)

- BMI ( $\geq 24 \text{ kg/m}^2$ ,  $\leq 24 \text{ kg/m}^2$ )
- Education level (elementary school and below, high school, university degree and postgraduate)
- Questionnaire with response and non-response subjects (if the subject performed ACQ and AQLQ at Visit 5 and had any questionnaire performed in each visit, the subject is defined as responder; otherwise, the subject is a non-response subject)
- Adherence (Good adherence or not)
- Patient expectation of asthma treatment
- Asthma severity class: Mild, Moderate, Severe (based on Patient Self-Assessment of Asthma Severity)
- Symptoms: Symptoms less than twice a month; Symptoms twice a month or more, but less than 4-5 days a week; Symptoms most days, or waking with asthma once a week or more; Daily symptoms, or waking with asthma once a week or more, and low lung function
- Hospital Type: PCCM, non-PCCM
- Geographic region: North, South
- ICS containing change: with-to-with, with-to-without, without-to-with, without-to-without ICS containing (From ICS containing to ICS containing, from ICS containing to no-ICS-containing, from no-ICS-containing to no-ICS-containing.)
- ICS-formoterol as reliever: with-to-with, with-to-without, without-to-with, without-to-without ICS-formoterol as reliever (From ICS-formoterol as reliever to ICS-formoterol as reliever, from ICS-formoterol as reliever, from no-ICS-formoterol as reliever, from no-ICS-formoterol as reliever, from no-ICS-formoterol as reliever.)
- Participants complete status: Missing at Week 24, not Missing at Week 24.
- Participants complete status: Missing at Week 48, not Missing at Week 48.

These analyses are exploratory and the result from these subgroup analyses will not affect the choice of the model for the primary analysis.

#### 5 INTERIM ANALYSIS

There will be two interim analyses, first interim analyses will mainly focus on the baseline when all subjects enrolled and finish baseline assessment, and the other will happen when all subjects complete week 12 visit.

First interim analysis includes the following parts:

- 1. Subject disposition
- 2. Demographics
- 3. Substance use nicotine
- 4. Asthma history
- 5. Historical asthma exacerbation
- 6. Prior and concomitant medications asthma/asthma related comorbidities
- 7. Prescribed medication asthma
- 8. ICS-based maintenance and/or reliever treatment
- 9. ACQ-5 average scores
- 10. Distribution of ACQ-5 average scores (Well controlled/Partly controlled/Not well-controlled) and its subgroup listed in Section 4.2.3.12
- 11. ICS-formoterol as reliever
- 12. Asthma treatment patterns
- 13. Numbers of severe asthma exacerbation
  - a. With ICS containing vs. without ICS containing
  - b. Good adherence vs. not
- 14. Health-related quality of life evaluated by Asthma Quality of Life Questionnaire for 12 years and older (AQLQ(S)+12) score
- 15. MARS-A average score
- 16. Hematology

- 17. Blood Gas
- 18. IgE
- 19. FeNO
- 20. Pulmonary Function Test (PFT)
- 21. Pulmonary Function Test-Post-BDT (PFT)

Second interim analysis includes the following parts:

- 1. Subject disposition
- 2. Demographics
- 3. Substance use nicotine
- 4. Asthma history
- 5. Historical asthma exacerbation
- 6. Prior and concomitant medications asthma/asthma related comorbidities
- 7. Prescribed medication asthma
- 8. ICS-based maintenance and/or reliever treatment
- 9. ACQ-5 average scores
- 10. Distribution of ACQ-5 average scores (Well controlled/Partly controlled/Not well-controlled) and its subgroup listed in Section 4.2.3.12
- 11. ICS-formoterol as reliever
- 12. Asthma treatment patterns
- 13. Patient evaluation on whose pulmonologists (whether their pulmonologists develop or review the written asthma action plan and watch the patient using their inhaler, checking their technique)
- 14. Numbers of severe asthma exacerbation
  - a. With ICS containing vs. without ICS containing
  - b. Good adherence vs. not

- 15. Health-related quality of life evaluated by Asthma Quality of Life Questionnaire for 12 years and older (AQLQ(S)+12) score
- 16. MARS-A average score
- 17. Inhaler skill score of subjects
- 18. Asthma knowledge score of subjects
- 19. Patient expectations of asthma treatment
- 20. Asthma knowledge questionnaire score of investigators
- 21. Adverse event
- 22. Hematology
- 23. IgE
- 24. FeNO
- 25. Pulmonary Function Test (PFT)
- 26. Pulmonary Function Test-Post-BDT (PFT)
- 27. Branchial Provocation Test

#### 6 REFERENCES

- FDA Guidance for Industry (issued July 2009) 'Drug-induced liver injury:
   Premarketing clinical evaluation':
   http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM174090.pdf
- 2. 中国医学装备协会呼吸病学专委会吸入治疗与呼吸康复学组,中国慢性阻塞性肺疾病联盟. 稳定期慢性气道疾病吸入装置规范应用中国专家共识[J]. 中华结核和呼吸杂志,2019,42(4):241-253.
- 3. Allen RM, Jones MP. The validity and reliability of an asthma knowledge questionnaire used in the evaluation of a group asthma education self-management program for adults with asthma. J Asthma. 1998;35(7):537-45.
- 4. 田庆秀,余丽君. 中文版支气管哮喘用药依从性量表的信效度检验[J]. 中华护理杂志,2014,49(5):621-624.
- 5. Mancuso CA, Rincon M, Robbins L, et al. Patients' expectations of asthma treatment. J Asthma. 2003 Dec;40(8):873-81.

## 7 APPENDIX

# 7.1 SAS sample code for proc GLIMMIX

```
proc GLIMMIX data=ics;

class visit (ref='0') hosp doct;

model mpd = visit /dist=binary link=logit oddsratio solution;

contrast 'week 48 vs baseline' time [1,4][-1,5];

random subjid hosp doct;

run;
```

# 7.2 SAS sample code for proc GENMODE

```
proc genmod data=ics;

class subjid hosp doct visit (ref='0')/ param=ref;

model mpd = visit / dist=bin link=logit;

repeated subject=subjid / corr=cs covb corrw;

run;
```

# 7.3 ASTHMA QUALITY OF LIFE QUESTIONNAIRE WITH STANDARDISED ACTIVITIES (AQLQ(S))

Self-administrated (≥12 years)

AstraZeneca 29-Jul-2024

| ASTHMA QUALITY OF LIFE QUESTIONNAIRE (S) | PATIENT ID: |
|------------------------------------------|-------------|
| SELF-ADMINISTERED | DATE: |

Please complete all questions by circling the number that best describes how you have been during the last 2 weeks as a result of your asthma.

HOW LIMITED HAVE YOU BEEN DURING THE LAST 2 WEEKS IN THESE ACTIVITIES AS A RESULT OF YOUR ASTHMA?

| | Totally<br>United | Extremely<br>Limited | Very<br>Limited | Moderate<br>Limitation | Some<br>Emitation | A Little<br>Limitation | Not at all<br>Limited |
|---|---|---|---|---|---|---|---|
| <ol> <li>STRENUOUS ACTIVITIES<br/>(such as hurrying, exercising,<br/>running up stairs, sports)</li> </ol> | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 2 MODERATE ACTIVITIES<br>(such as waking, housework,<br>gardening, shopping, climbing<br>stairs) | 1 | 2 | 3 | 4. | 5 | 6 | 7 |
| <ol> <li>SOCIAL ACTIVITIES<br/>(such as talking, playing with<br/>pets/children, visiting<br/>friends/relatives)</li> </ol> | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| WORK/SCHOOL-RELATED<br>ACTIVITIES* (lasks you have<br>to do at work/in school) | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 5. SLEEPING | 1 | 2 | 3 | 4 | 5 | 6 | 7 |

<sup>&</sup>quot;If you are not employed or self-employed, these should be tasks you have to do most days.

#### HOW MUCH DISCOMFORT OR DISTRESS HAVE YOU FELT DURING THE LAST 2 WEEKS?

| | A Very<br>Great Deal | A Grant<br>Deal | A Good<br>Dear | Moderate<br>Amount | Some | Very<br>Little | None |
|---|---|---|---|---|---|---|---|
| How much discomfort or distress have you felt over the last 2 weeks as a result of CHEST TIGHTNESS? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |

Mcd-fied September 2010 AOLO(S) 212 years SA North American English Version

# STATISTICAL ANALYSIS PLAN D589BC00027 - ed.4.0

| | | ESTIONNA | ٠. | | ATIENT IC | | | - |
|---|---|---|---|---|---|---|---|---|
| ELF | -ADMINISTERED | | | D | ATE: | | | |
| 1 GE | NERAL, HOW MUCH OF THE | TIME DUR | ING THE | LAST 2 W | EEKS DID | YOU: | | |
| | | All of<br>the Time | Most of<br>the Time | A Good<br>Bit of the<br>Time | Some of the Time | A Late of<br>the Time | Hardly Any<br>of the Tene | None of<br>the Time |
| 7. | Feel CONCERNED ABOUT HAVING ASTHMA? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 8 | Feet SHORT OF BREATH as a result of your asthma? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 9. | Experience asthma<br>symptoms as a RESULT<br>OF BEING EXPOSED TO<br>CIGARETTE SMOKE? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 10. | Experience a WHEEZE in your chest? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 11. | Feel you had to AVOID A<br>SITUATION OR<br>ENVIRONMENT BECAUSE<br>OF CIGARETTE SMOKE? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| ΟW | MUCH DISCOMFORT OR DIS | TRES\$ HA | VE YOU | FELT DUR | ING THE | LAST 2 WI | EEKS? | |
| | | A Very<br>Great Deal | A Great<br>Dost | A Good<br>Deal | Moderate<br>Amount | \$ome | Very<br>Little | None |
| 12. | How much discomfort or distress have you felt over the last 2 weeks as a result of COUGHING? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| | distress have you felt over<br>the last 2 weeks as a result | · | _ | - | · | · | 6 | 7 |
| | distress have you felt over<br>the last 2 weeks as a result<br>of COUGHING? | · | _ | - | · | · | 6<br>Hardy Any<br>of the Time | 7<br>None of<br>the Time |
| I GE | distress have you felt over<br>the last 2 weeks as a result<br>of COUGHING? | TIME DUR | LING THE | LAST 2 W | EEKS DID | YOU: | Hardy Any | Nane of |

Modified September 2010 AOLO(S) 212 years SA North American English Version

# STATISTICAL ANALYSIS PLAN D589BC00027 - ed.4.0

PATIENT ID: ASTHMA QUALITY OF LIFE QUESTIONNAIRE (S) DATE:  SELF-ADMINISTERED

IN GENERAL, HOW MUCH OF THE TIME DURING THE LAST 2 WEEKS DID YOU:

| | | All of<br>the Time | Most of<br>the Tyme | A Good<br>Ba of the<br>Time | Some of<br>the Time | A Little of<br>the Time | Hardly Any<br>of the Time | None of<br>the Time |
|---|---|---|---|---|---|---|---|---|
| 15. | Feel CONCERNED ABOUT<br>THE NEED TO USE<br>MEDICATION for your<br>asthma? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 16. | Feel the need to CLEAR<br>YOUR THROAT? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 17. | Experience asthma<br>symptoms as a RESULT OF<br>BEING EXPOSED TO<br>DUST? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 18. | Experience DIFFICULTY<br>BREATHING OUT as a<br>result of your asthma? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 19. | Feel you had to AVOID A<br>SITUATION OR<br>ENVIRONMENT BECAUSE<br>OF DUST? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 20. | WAKE UP IN THE<br>MORNING WITH ASTHMA<br>SYMPTOMS? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 21. | Feel AFRAID OF NOT<br>HAVING YOUR ASTHMA<br>MEDICATION AVAILABLE? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 22. | Feel bothered by HEAVY<br>BREATHING? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 23. | Experience asthma symptoms as a RESULT OF THE WEATHER OR AIR POLLUTION OUTSIDE? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 24. | Were you WOKEN AT<br>NIGHT by your asthma? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 25. | AVOID OR LIMIT GOING<br>OUTSIDE BECAUSE OF<br>THE WEATHER OR AIR<br>POLLUTION? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |

Modified September 2010 AQLQ(S) ≥12 years SA North American English Version

# STATISTICAL ANALYSIS PLAN D589BC00027 - ed.4.0

| AST | ASTHMA QUALITY OF LIFE QUESTIONNAIRE (S | | IAIRE (S) | P/ | PATIENT ID: | | | |
|---|---|---|---|---|---|---|---|---|
| SELF | -ADMINISTERED | | | D/ | ATE: | | | |
| IN GE | NERAL, HOW MUCH OF THE | NME DU | RING THE | LAST 2 W | EEK\$ DI | YOU: | | <del></del> |
| | | All of<br>the Time | Most of<br>the Time | A Good<br>Bit of the<br>Time | Some of<br>the Time | A Little of<br>the Time | Hardy Any<br>of the Time | None of<br>the Time |
| 26. | Experience asthma<br>symptoms as a RESULT OF<br>BEING EXPOSED TO<br>STRONG SMELLS OR<br>PERFUME? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 27. | Feel AFRAID OF GETTING<br>OUT OF BREATH? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 28 | Fool you had to AVOID A<br>SITUATION OR<br>ENVIRONMENT BECAUSE<br>OF STRONG SMELLS OR<br>PERFUME? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 29. | Has your asthma<br>INTERFERED WITH<br>GETTING A GOOD NIGHT'S<br>SLEEP? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| 30. | Have a feeling of FIGHTING FOR AIR? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| HOW | LIMITED HAVE YOU BEEN DU | RING TH | RE LAST 21 | WEEKS? | | | | |
| | | Severally<br>Limited<br>Most Not<br>Done | Very Limited | Moderately<br>Limited<br>Several Not<br>Done | Sighty<br>Limited | Very Slight:<br>Limited<br>Very Few No<br>Done | Limned At A | Not Limited<br>Have Done<br>All Activities |
| 31 | Think of the OVERALL RANGE OF ACTIVITIES that you would have liked to have done during the last 2 weeks. How much has your range of activities been limited by your asthma? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |

Modified September 2010 AQLQ(S) ≥12 years SA North American English Version

# STATISTICAL ANALYSIS PLAN D589BC00027 – ed.4.0

AstraZeneca 29-Jul-2024

| ASTHMA QUALITY OF LIFE QUESTIONNAIRE (S) | | P | ATIENT ID | ); | | | |
|---|---|---|---|---|---|---|---|
| SELF-ADMINISTERED | ELF-ADMINISTERED | | D | ATE: | | | |
| HOW LIMITED HAVE YOU BEEN DU | URING TH | E LAST 21 | WEEKS? | | | | |
| | Totally<br>Limited | Extremely<br>Limited | Very<br>Limited | Moderate<br>Limitation | Some<br>Limitation | À Little<br>Limitation | Not at as<br>Limited |
| 32. Overall, among ALL THE<br>ACTIVITIES that you have<br>done during the last 2 weeks,<br>how limited have you been by<br>your asthma? | 1 | 2 | 3 | 4 | 5 | 6 | 7 |

#### DOMAIN CODE:

Symptoms: 6, 8, 10, 12, 14, 18, 18, 20, 22, 24, 29, 30 Activity Limitation: 1, 2, 3, 4, 5, 11, 19, 25, 28, 31, 32 Emotional Function: 7, 13, 15, 21, 27 Environmental Stimuli: 9, 17, 23, 26

Modified September 2010 AQLQ(S) ≥12 years SA North American English Version